CLINICAL TRIAL: NCT01350648
Title: The Natural History of Liver Disease in a Cohort of Participants With Hepatitis B and/or Hepatitis C With or Without HIV Infection
Brief Title: Long-Term Study of Liver Disease in People With Hepatitis B and/or Hepatitis C With or Without HIV Infection
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 110152; 11-CC-0152
Record Dates: First submitted 2011-05-07; First posted 2011-05-10 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis B; Hepatitis C; HIV-HCV Co-Infection
Keywords: Viral Hepatitis; Acquired Immunodeficiency Syndrome (AIDS); Hepatocellular Carcinoma; HIV-HCV Co-Infection; Liver Neoplasms; Natural History
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Acquired Immunodeficiency Syndrome; Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- HBV and HCV Co-infection: HBV and HCV Co-infection
- Hepatitis B: Hepatitis B alone
- Hepatitis C: Hepatitis C alone
- HIV and HBV and HCV Tri-Infection: HIV and HBV and HCV Tri-Infection
- HIV and HBV Co-infection: HIV and HBV Co-infection
- HIV/HCV Co-Infection: HIV and HCV Co-infection

SUMMARY:
Background:

- Hepatitis B and hepatitis C can cause liver damage. They can also cause serious illness, including liver cancer, and even death. This study will follow people who have hepatitis B or hepatitis C. The purpose is to understand more about how these viruses affect the immune system over the long term (up to 10 years). The study will also compare how these viruses affect people who do and do not have HIV, the virus that causes AIDS.

Objectives:

* To do a long-term study of hepatitis B and hepatitis C infection.
* To study the effects of hepatitis B and hepatitis C infection in people do and do not have HIV.

Eligibility:

- People at least 18 years of age who have hepatitis B or hepatitis C and have a regular doctor for their medical care.

Design:

* Participants will be screened with a physical exam and medical history. Those who do not have a regular doctor to provide medical care during the study will not be able to take part.
* Participants will have yearly visits with study researchers for up to 10 years. These tests will be done at each visit.
* Medical history and physical exam.
* Questionnaire (optional) on emotions, sexual behaviors, use of alcohol and drugs, and quality of life.
* Blood and urine tests, including HIV testing.
* Tissue sample collections for those who have had a liver or other tissue biopsy.
* Participants may leave the study at any time. They will receive the standard of care from their regular doctor throughout the study.

DETAILED DESCRIPTION:
Chronic viral hepatitis is a major health problem affecting millions globally. The immunosuppressed population, especially those with HIV infection, remains at particular risk and the incidence of hepatocellular carcinoma (HCC) is increasing in the US and worldwide, with high rates in those who are cirrhotic, and is the 10th most common cause of death in the US.

HIV-hepatitis coinfection is problematic in that HIV patients are currently living longer on highly active antiretroviral therapy (HAART). Those who are coinfected with HBV and/or HCV progress more rapidly to cirrhosis and hepatic failure. Further research on the epidemiology, optimal screening and new therapeutic approaches in persons with advanced liver disease, in the setting of effective treatment for viral hepatitis is needed.

The primary objective of the proposed study is to characterize viral liver disease and factors affecting the natural history of viral liver disease in persons with and without HIV with an emphasis on those living in the Washington DC metropolitan area. The cohort will be designed to study research questions with respect to liver disease, disease pathogenesis using genomics, proteomics, and immunologic disease models. Secondary objectives include study of the immunopathogenesis of HBV and HCV disease progression in HIV infected subjects. In addition, this is an invaluable opportunity to determine the prevalence and risk factors associated with the development of hepatocellular carcinoma, the longterm effects of HCV clearance with DAAs, along with biomarker profile(s) for diagnosis and outcome. Moreover, this will serve as a catchment protocol to select appropriate participants for novel HBV and HCV therapeutic trials.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for participation on this protocol, a participant must satisfy all of the following conditions:

1. Be greater than or equal to 18 years old
2. HBV-infected and/or HCV-infected, or was HCV-infected and successfully treated
3. Willing to undergo genetic testing
4. Willingness to allow study staff to review your medical records between research visits
5. Willing to have samples stored for future research
6. Must have an identifiable primary care physician
7. Willing to undergo HIV testing
8. Childbearing female must test negative for pregnancy

An HBV infected individual is defined as any individual with documentation of the following:

- Positive Hepatitis B surface antigen within the past 12 months or HBV DNA positive, or prior documentation if the individual is currently on active therapy

An HCV infected individual is defined as any individual with documentation of the following in the past:

- Positive HCV antibody and/or positive HCV RNA test (HCV RNA of 2,000 IU/mL or greater)

An HIV infected individual is defined as any individual with documentation of the following:

- Positive Enzyme Linked Immunosorbent Assay followed by a positive Western Blot or detectable HIV viral load or HIV viral less than 50 copies/mL with documentation this individuals is curently on an active HIV antiretroviral regimen.

EXCLUSION CRITERIA:

A participant will be ineligible to participate on this study if any of the following criteria are met:

1. Unable to comply with research study visits
2. Poor venous access
3. Have any condition that the investigator considers a contraindication to study participation.
4. Childbearing female with positive pregnancy test

Co-enrollment Guidelines: Participants may be enrolled in other protocols as long as the amount of research blood drawn does not exceed the acceptable NIH guidelines.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NIH NIAID Outpatient Clinic 8 Participants, local Washington DC Primary Clinics, and formerly the Washington DC VA Clnic
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2011-08-23 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Progression of liver disease in patients with HCV | Annual visits
  Exams and labs
Progression of liver disease in patients with HBV | Annual visits
  exam and labs

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - VA Medical Center, Washington D.C., Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. Hepatology. 2009 Sep;50(3):661-2. doi: 10.1002/hep.23190. No abstract available. PMID 19714720
- [Background] Lavanchy D. Hepatitis B virus epidemiology, disease burden, treatment, and current and emerging prevention and control measures. J Viral Hepat. 2004 Mar;11(2):97-107. doi: 10.1046/j.1365-2893.2003.00487.x. PMID 14996343
- [Background] Alter MJ. Epidemiology of viral hepatitis and HIV co-infection. J Hepatol. 2006;44(1 Suppl):S6-9. doi: 10.1016/j.jhep.2005.11.004. Epub 2005 Nov 21. PMID 16352363
- [Derived] Balmaceda JB, Aepfelbacher J, Belliveau O, Chaudhury CS, Chairez C, McLaughlin M, Silk R, Gross C, Kattakuzhy S, Rosenthal E, Kottilil S, Kleiner DE, Hadigan C. Long-term changes in hepatic fibrosis following hepatitis C viral clearance in patients with and without HIV. Antivir Ther. 2019;24(4):451-457. doi: 10.3851/IMP3327. PMID 31359874
- [Derived] Chaudhury CS, Mee T, Chairez C, McLaughlin M, Silk R, Gross C, Kattakuzhy S, Rosenthal E, Kottilil S, Stanley TL, Hadigan C. Testosterone in Men With Chronic Hepatitis C Infection and After Hepatitis C Viral Clearance. Clin Infect Dis. 2019 Aug 1;69(4):571-576. doi: 10.1093/cid/ciy965. PMID 30715229
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-CC-0152.html